CLINICAL TRIAL: NCT00050726
Title: Substudies of ESPRIT: ESPRIT Influenza Vaccine Substudy (FLUVAC) and ESPRIT Tetanus-Pneumococcal Vaccine Substudy (TEPVAC)
Brief Title: Studies of Influenza Vaccine and Tetanus-Pneumococcal Vaccine in HIV-infected Patients Receiving Interleukin-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: DAIDS, NIAID
Purpose: Treatment
Other Study IDs: 010171; 01-I-0171
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Immunotherapy; HIV; IL-2
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2

SUMMARY:
This investigation is a sub-study of the 6-year multinational ESPRIT (Evaluation of Subcutaneous Proleukin in a Randomized International Trial) protocol. It will compare the effectiveness of the influenza (FLUVAC) and tetanus-pneumococcal (TEPVAC) vaccines in HIV-infected patients receiving interleukin-2 (IL-2) plus anti-HIV drugs with those receiving only anti-HIV drugs. IL-2 is a protein naturally produced by immune cells called lymphocytes. Lymphocytes from patients with HIV do not produce IL-2 normally. The ESPRIT trial is evaluating whether HIV-infected patients treated with antiretroviral drugs plus IL-2 have fewer serious infections and improved survival than those receiving only anti-HIV drugs.

Participants in this sub-study will be drawn from patients enrolled in ESPRIT. They must be 18 years of age or older, have HIV infection with no symptoms of significant HIV illness. They will be vaccinated against either influenza or tetanus and pneumococcus, as follows:

FLUVAC

Potentially eligible patients will be screened for the FLUVAC study during an ESPRIT follow-up visit. Those who are eligible and agree to participate will have 10 ml (1 tablespoon) of blood drawn to assess baseline antibody levels and then receive the vaccination. They will be vaccinated annually for 3 years. A blood sample (10 ml) will be drawn 1 month after each vaccination to measure the immune response. Some of the blood drawn for this study will be stored and used for research purposes.

TEPVAC

Participants will have 10 ml of blood drawn to assess their baseline antibody levels. They will receive two vaccinations (tetanus and pneumococcus) 12 months after enrolling in ESPRIT and another two vaccinations 24 months after enrollment. A blood sample (10 ml) will be drawn 1 month after each vaccination to measure the immune response. Some of the blood drawn for this study will be stored and used for research purposes.

DETAILED DESCRIPTION:
Evaluation of Subcutaneous Proleukin in a Randomized International Trial (ESPRIT) is a 4,000 patient, 6-year study investigating the clinical effect of interleukin-2 (IL-2) in patients with HIV infection. Because of the size and duration of this study, substudies to the parent trial are being performed in order to improve the knowledge regarding the use of IL-2 in HIV-infected individuals and to enhance the overall scientific output of this international effort. This protocol will serve as the umbrella under which the ESPRIT substudies will be performed at the National Institutes of Health Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA - ESPRIT PROTOCOL:

Documentation of HIV-1 infection by any licensed ELISA test and confirmed by a second method (e.g. Western Blot); or any one of the following at any time: detectable HIV p24 antigen, quantifiable plasma HIV RNA, or detectable proviral DNA.

Absolute CD4 plus cell count of greater than or equal to 300/mm(3) within 45 days prior to randomization. (For patients who are status post-splenectomy, also a CD4 plus cell percentage greater than or equal to 20%.)

No evidence of active clinical disease for at least one year, in the judgement of the clinician, for any AIDS-defining illness (category C., CDC, 1993) or any of the following conditions: extrapulmonary Pneumocystis carinii disease; multi-dermatomal Herpes zoster (greater than or equal to 10 lesions in a non-contiguous site); American trypanosomiasis (Chagas disease) of the CNS; Penicillium marneffii disease; visceral leishmaniasis; non-Hodgkin's lymphoma of any cell-type; Hodgkin's lymphoma; bartonellosis; microsporidiosis (greater than 1 month's duration); nocardiosis; invasive aspergillosis; or Rhodococcus equi disease.

Age greater than or equal to 18 years.

Laboratory values (within 45 days prior to randomization):

AST or ALT less than or equal to 5 x the upper limit of normal (ULN).

Total or direct bilirubin less than 2 x ULN (Patients with hyperbilirubinemia due to Gilbert's syndrome or indinavir therapy may have a serum bilirubin up to 5 x ULN.)

Creatinine less than or equal to 2.0 mg/dl (177 micro mol/L).

Platelet count greater than or equal to 50,000/mm(3).

On or initiating combination antiretroviral therapy at the time of randomization. Antiretroviral therapy can include agents (approved and investigational) administered through routine care or through participation in clinical trials or expanded access programs.

Signed informed consent form.

INCLUSION CRITERIA - FLUVAC STUDY:

Patients eligible for the ESPRIT trial are eligible for the FLUVAC study, except for patients with known allergy to egg, a history of allergic reaction(s) to influenza vaccination or who had an influenza vaccine less than or equal to 6 months after ESPRIT randomization and during the influenza vaccine season, i.e. between September 1st and January 31st on the Northern hemisphere and between February 1st and June 30th on the Southern hemisphere.

The inclusion criteria will be the same as the ESPRIT protocol.

EXCLUSION CRITERIA - ESPRIT PROTOCOL:

Prior rIL-2 therapy.

Concurrent malignancy requiring cytotoxic chemotherapy.

Use of systemic corticosteroids, immunosuppressants, or cytotoxic agents within 45 days prior to study randomization.

Any CNS abnormality that requires ongoing treatment with antiseizure medication.

Current or historical autoimmune/Inflammatory diseases including: Inflammatory bowel disease (Chron's disease, ulcerative colitis); Psoriasis; Optic neuritis; or Any autoimmune/inflammatory diseases with potentially life-threatening complications.

Pregnancy (For women of childbearing potential, a negative pregnancy test, serum or urine, is required within 14 days prior to randomization.)

Breast feeding.

EXCLUSION CRITERIA - FLUVAC:

As for the ESPRIT protocol with the addition patients allergic to egg, with a history of allergic reaction(s) to influenza vaccination or who had a influenza vaccine less than or equal to 6 months before inclusion are not eligible for this study.

EXCLUSION CRITERIA - TEPVAC:

As for the ESPRIT protocol with the additions of patients with a history of allergic reaction to the study vaccines and/or a planned (or given) vaccination with either of the study vaccines within the 12 months following ESPRIT randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620
Dates: Start 2001-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with eroconversion to one or more vaccine antigens. | Month1 post-vaccination.

CONTACTS AND LOCATIONS:
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Hvidovre University Hospital@@@Copenhagen, Denmark, Copenhagen, Denmark

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2001-I-0171.html